CLINICAL TRIAL: NCT00219752
Title: Phase II Trial to Study the Tolerability and the Effectiveness of Imatinib in Patients With Chronic Myelogenous Leukemia in Chronic Phase With Age More Than 70, Diagnosis of CML is Being Performed Within 1 Year
Brief Title: Safety and Efficacy of Imatinib in Chronic Myelogenous Patients Older Than 70 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020948; CSTI571AFR04
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2005-12-22 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CML - ederly patients - Imatinib mesylate
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib mesylate 400 mg

SUMMARY:
The aim of this phase II trial is asses the tolerability and the effectiveness of imatinib in patients with chronic myelogenous leukemia in chronic phase with age more than 70, diagnosis of cml is being performed within 1 year. Quality of life will be carefully assessed.

DETAILED DESCRIPTION:
Patients will received Imatinib at a dose of 400mg daily. Tolerability and quality of life will be assessed Secondary objectives are : to evaluate the survival without progression, the survival without event, the overall survival, the hematologic, cytogenetic and molecular responses at various check points.

Duration of responses and failure to respond will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* CML Ph+ (assessed by cytogenetic or FISH)
* Chronic phase with less than 5% bone marrow blasts
* Diagnosis within 12 months
* Age ≥ 70 year at inclusion
* PS grade 0 to 2 (ECOG)
* Mini mental status more than 25
* Hydroxyurea optional before Imatinib
* Adequate end organ function, defined as the following: total bilirubin <1.5x uln, sgpt <3x uln, creatinine <1.5x uln.

Exclusion Criteria:

* patients who cannot sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of the hospital
* Mini mental status ≤ 25
* patients who are not able to adequately take the study drug
* Age less than 70 y
* accelerated or blastic phase
* previous therapy with imatinib or interferon
* HIV positivity

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30
Dates: Start 2002-05; Study Completion 2007-05

PRIMARY OUTCOMES:
Tolerability
Quality of life

SECONDARY OUTCOMES:
. the survival without progression
. the survival without event
. the overall survival
. the hematologic cytogenetic and molecular responses at various check points.
. duration of responses and failure to respond

CONTACTS AND LOCATIONS:
Overall Officials: François GUILHOT, MD, Study Chair — Department of Oncology hematology and Cell therapy, University Hospital , 86021 Poitiers - FRANCE; Philippe ROUSSELOT, MD, Principal Investigator — Department of Hematology and Oncology - University Hospital "Saint Louis" - 75475 PARIS cedex 10 (FRANCE)
Locations (1):
- University Hospital, Poitiers, France